CLINICAL TRIAL: NCT00353626
Title: Gait Evaluation of Experienced Post Traumatic Below Knee Amputees
Brief Title: Gait Evaluation of Experienced Below Knee Amputees
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Uri Givon MD, Sheba Medical Center
Other Study IDs: SHEBA-06-4211-UG-CTIL
Record Dates: First submitted 2006-07-16; First posted 2006-07-18 (Estimated); Last update posted 2008-03-24 (Estimated); Status verified 2008-03

CONDITIONS: Amputations, Traumatic
Keywords: Amputation; trans tibial; prosthesis; motion analysis
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Post traumatic amputees with an experience of over 3 months of prosthesis use at home, without any known difficulty using the prosthesis and without stump pathology, using no assistive devices, will be examined in a 3 D computerized gait laboratory. Kinematic and kinetic parameters of gait will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Post traumatic trans tibial amputees
* No stump pathology
* No assistive devices
* No technical difficulty

Exclusion Criteria:

* Vascular or DM background
* Stump pathology
* Gait difficulties
* Assistive device

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Trans tibial amputees without pain or complaints about stump or prosthesis,using their prosthesis more than 3 months.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2006-06; Primary Completion 2007-07 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uri Givon, MD, Principal Investigator — Motion analysis Laboratory, Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel